CLINICAL TRIAL: NCT05593848
Title: Comparative Study of the Effects of Intratissue Percutaneous Electrolysis vs. Dry Needling in the Treatment of Myofascial Pain Syndrome in Subjects With Non-specific Shoulder Pain
Brief Title: Intratissue Percutaneous Electrolysis vs Dry Needling in Myofascial Pain Syndrome of Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Roberto Méndez Sánchez, Professor, PhD, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 419-2019 USalamanca
Record Dates: First submitted 2022-10-19; First posted 2022-10-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Shoulder Pain; Myofascial Pain Syndrome
Keywords: Intratissue Percutaneous Electrolysis; Dry Needling; Myofascial trigger points; infraspinatus muscle; non-specific shoulder pain
MeSH Terms: conditions — Shoulder Pain; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Intratissue Percutaneous Electrolysis Group) (Experimental): The treatment to be performed in the Intratissue percutaneus electrolysis Group will consist of:
  1. Palpation and localization of the myofascial trigger points in the infraspinatus muscle of the affected shoulder.
  2. Application of the ultrasound-guided intratissue percutaneus electroysis technique (1 or 2 approaches) on the myofascial trigger points with the greatest clinical manifestations for the subject. The needle will remain at intramuscular level without movement and a galvanic current discharge will be applied in the area, through the needle, whose intensity will oscillate between 0.5 and 3 milliAmperes (mA).
  3. Performance of an eccentric work protocol of the infraspinatus muscle to reduce post-puncture pain.
  Interventions: Procedure: Intratissue Percutaneous Electrolysis
- Active Control Group (Dry Needling Group) (Active Comparator): The treatment to be performed in the Dry Needling Group will consist of:
  1. palpation and localization of myofascial trigger points in the infraspinatus muscle of the affected shoulder.
  2. Application of the ultrasound-guided dry needling technique (1 or 2 approaches) on the myofascial trigger points with major clinical manifestations for the subject. The physiotherapist will move the needle into the muscle using Hong's rapid entry and exit technique.
  3. Performance of an eccentric work protocol of the infraspinatus muscle to reduce post-puncture pain.
  Interventions: Procedure: Dry Needling

INTERVENTIONS:
Procedure: Intratissue Percutaneous Electrolysis — Each subject will undergo 3 treatment sessions spaced one week apart. Ultrasound-guided Intratissue Percutaneous Electrolysis in the myofascial trigger points of the infraspinatus muscle
  Arms: Experimental Group (Intratissue Percutaneous Electrolysis Group)
Procedure: Dry Needling — Each subject will undergo 3 treatment sessions spaced one week apart. Ultrasound-guided dry needling in the myofascial trigger points of the infraspinatus muscle
  Arms: Active Control Group (Dry Needling Group)

SUMMARY:
This is a parallel-group randomised clinical trial:

Primary purpose: To analyse the clinical changes produced by two different physiotherapy treatments (Intratissue Percutaneous Electrolysis and Dry Needling) for myofascial trigger points in the infraspinatus muscle in subjects with non-specific shoulder pain.

Hypothesis: A physiotherapy treatment including Intratissue Percutaneous Electrolysis therapy present greater benefits in terms of pain reduction and increased mobility and functionality rather than Dry Needling treatment in subjects with non-specific shoulder pain.

The intervention consisted of 3 treatment sessions, different according to the group, once a week. Seven evaluation points were performed, two pre-intervention evaluations one week apart and after the second one the first treatment session was performed. The third and fourth assessments were prior to the second and third treatment sessions, one week apart. The fifth, sixth and seventh assessments were conducted one week, one month and two months after the last treatment session in each group.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients suffering from shoulder pain during at least three months before intervention protocol starts.
* Patients with free passive range of movement and at least 15 degrees active external rotation in the affected shoulder.
* Patients willing to participate in the study and return for all scheduled follow-up visits.
* Patient is capable of giving, and has given, written informed consent.

Exclusion Criteria:

* Patients with a previous medical diagnosis (tendon rupture, bursitis, etc.) or a traumatic history that justifies shoulder pain.
* Patients with unstable or uncontrolled angina, uncontrolled heart failure, or serious uncontrolled ventricular arrhythmias.
* Patients allergic to metal or those who have needle phobia.
* Patient that has participated in any other shoulder pain treatment research study within 30 days prior.
* Patients that had prior shoulder surgery.
* Patients that are currently being treated with a narcotic or NSAIDs and/or has used analgesics or NSAIDs within the 72 hours prior.
* Patients that has a known bleeding disorder or that are currently being treated with anticoagulant therapy.
* Pregnant women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain intensity, before, during and after the intervention | 4 months (7 points)
  Numerical pain rating scale (score 0-10 points)

SECONDARY OUTCOMES:
Changes in Shoulder flexion range of motion, before, during and after the intervention | 4 months (7 points)
  The range of motion in flexion will be measured with an inclinometer to assess changes in the mobility to shoulder pain subjects
Changes in Shoulder external rotation range of motion, before, during and after the intervention | 4 months (7 points)
  The range of motion in external rotation will be measured with an inclinometer to assess changes in the mobility to shoulder pain subjects
Changes in Pressure pain threshold at proximal myofascial trigger point of the infraspinatus muscle, before, during and after the intervention | 4 months (7 points)
  The pressure threshold will be recorded using a digital algometer.
Changes in Pressure pain threshold at distal myofascial trigger point of the infraspinatus muscle, before, during and after the intervention | 4 months (7 points)
  The pressure threshold will be recorded using a digital algometer (Pain Test™ FPIX 10)
Changes in Strength in shoulder external rotation before, during and after the intervention | 4 months (7 points)
  The strength will be recorded with wireless MicroFET 2: Hand-held dynamometer for force assessment.
Changes in Hand grip strength, before, during and after the intervention | 4 months (7 points)
  The strength will be recorded with Jamar Plus: Digital dynamometer to assess grip strength.
Changes in Disability and functionality of the upper limb, before, during and after the intervention | 4 months (7 points)
  To measure the upper limb disability and functionality we will use the Disabilities of the Arm, Shoulder and Hand (DASH), which is a validated questionnaire that measures the functionality and disability that shoulder pain generates in the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Méndez-Sánchez, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Spain